CLINICAL TRIAL: NCT04751305
Title: The Feasibility of a Remote Maintenance Exercise Program for Cancer Survivors Supported by Health Coaching.
Brief Title: Remote Exercise Maintenance With Health Coaching for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREBA.CC-19-0206
Record Dates: First submitted 2021-01-13; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-12

CONDITIONS: Cancer Survivors
Keywords: mHealth; Health Coaching; Exercise; Online delivery
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: At the beginning of the remote ACE maintenance program participants are randomized into either the exercise only group or the exercise with additional health coaching group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The certified exercise physiologists (CEP) instructing the exercise classes were unaware of the intervention each participant was assigned to. The CEP administering the physical functioning assessment was unaware of the participants intervention and was not the participants exercise class instructor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACE Remote Maintenance Program with Health Coaching (Experimental): The participants received online delivered (over zoom) group based exercise classes (2x/wk for first 2 weeks; 1x/wk for the remaining weeks) followed by a 15 minute post workout social session. Participants also received a PDF of a home-based exercise program with embedded videos and a Garmin Vivosmart4 activity tracker. The accelerometer is not intended to be an active part of the intervention but is used to gather an objective measure of PA levels. Additionally, the health coaching intervention received weekly zoom calls that were focused on being participant-centered, built on a coach participant relationship, and included participant-determined goals, a self-discovery process to find solutions, patient accountability, and education.
  Interventions: Behavioral: Health Coaching; Behavioral: Online delivered Exercise Classes
- Only ACE Remote Maintenance Program (Active Comparator): The participants received online delivered (over zoom) group based exercise classes (2x/wk for first 2 weeks; 1x/wk for the remaining weeks) followed by a 15 minute post workout social session. Participants also participants received a PDF of a home-based exercise program with embedded videos and a Garmin Vivosmart4 activity tracker. The accelerometer is not intended to be an active part of the intervention but is used to gather an objective measure of PA levels.
  Interventions: Behavioral: Online delivered Exercise Classes

INTERVENTIONS:
Behavioral: Health Coaching — The weekly health coaching (HC) calls were structured to be participant-centered, built on a coach participant relationship, and include participant-determined goals, a self-discovery process to find solutions, patient accountability, and education. Before each HC call, the participants received a short questionnaire on fatigue, QOL, stress, loneliness, and social support which enabled tailoring the HC call to the individual. Educational topics are discussed in the following order: Goal Setting, Monitoring Behaviour, Barrier Management, Social Support, Stress Management, Adapting the Program, Self-Compassion, Sleep & Nutrition, Reflection, Health Media, Remote Resources, and Maintaining Motivation. However, the order of the educational topics can be adjusted based on the specific participants' needs each week. At the half-way point of the intervention, the participant provided feedback on the HC calls, ensuring optimization of HC impact.
  Arms: ACE Remote Maintenance Program with Health Coaching
Behavioral: Online delivered Exercise Classes — The group based remote exercise program was delivered over the Zoom application (2x/wk for first 2 weeks; 1x/wk for the remaining weeks). Classes were one hour long with a ten minute warm up, 40 minute strength and conditioning focused exercise circuits, and a ten minute stretch. Each class was followed by additional time to provide participants with an opportunity to interact with each other, fostering social support.

SUMMARY:
The feasibility of an online maintenance exercise program for cancer survivors supported by health coaching.

DETAILED DESCRIPTION:
Purpose: The primary aim of this proposed mixed-methods study is to determine the feasibility of implementing a home-based exercise program with the support of telephone-based health coaching (HC). The secondary aim is to test the effectiveness of the program on physical activity (PA) levels, psychosocial well-being, and physical functioning.

Background: Cancer is the leading cause of death in Canada, and one in two Canadians will be diagnosed with cancer in their lifetime. Cancer treatments can prolong life, however it is often at the expense of a multitude of negative symptoms and side-effects that diminish quality of life (QOL). Exercise is one of the most effective and safe options among non-pharmaceutical interventions to manage the psychological and physiological side effects of cancer. Despite the known benefits, PA levels amongst cancer survivors are low. The main barriers to exercise in cancer survivors include lack of time, treatment-related side effects, and fatigue. One factor used to address these potential barriers is to have flexibility in programming, including varying sites for delivery of programs (centre vs home). While there is a preference towards home-based programs, adherence and maintenance rates are generally lower compared to group-based programs.

Rationale: Home-based programs can address the preferences of cancer survivors and potential barriers of exercise, such as access and lack of time. However, there is a need to increase adherence in a home-based program setting.

Objectives/ Research Question: The primary outcome measure of this pilot study is feasibility, while the secondary outcome measures include PA levels, physical functioning, and patient reported outcomes (PRO). We hypothesize that a home-based exercise program, designed to promote self-efficacy and supported by HC, will be maintained, and will improve physical activity levels, self-efficacy in managing the additional burden of isolation, and symptom management, such as chronic fatigue and QOL. The data collected will be used to inform the implementation of a home-based maintenance exercise program.

Research Plan: Assessments of the two intervention arms 1) online group maintenance classes (tapered sessions, 2x/wk for first 2 weeks; 1x/wk for remaining 6 weeks); and 2) online group maintenance classes (same tapered format) with HC (1x/week for approximately 30 minutes) will occur at baseline and post intervention. The first wave of the intervention was run from May until July 2020 for 8 weeks and the second wave was run from September until December 2020 for 12 weeks. Feasibility is the primary outcome measure, including recruitment rate (% who participate from those eligible), assessment completion, safety (adverse event reporting), attendance to remote maintenance classes, HC call completion, and attrition rates. Secondary outcomes include PROs of fatigue, loneliness, stress, social support, self-efficacy, QOL, and PA levels; and measures of physical functioning. Fatigue will be assessed using the FACIT-F. Social support will be assessed through the OSSS-3. Stress and loneliness will be assessed with the PSS and ULS-6 respectively. Self-efficacy will be assessed with a modified barrier SE scale and QOL with the FACT-general questionnaire. PA levels will be monitored objectively through weekly PA levels recorded with an accelerometer, and pre-/post intervention with the self-reported GLTEQ. Physical functioning assessments will be conducted remotely with a clinical exercise physiologist. Semi-structured interviews conducted post-intervention will focus on feasibility, including participant satisfaction, barrier management, pros/cons to the home-setting, value of the health coaching support, and facilitators to maintaining PA levels.

Significance: Exercise improves physical and psychological symptom burden from cancer treatment and enhances QOL. During COVID necessitated social isolation, a feasible and effective home-based exercise program may increase the capacity of cancer survivors to engage in regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Diagnosed with Cancer within the last 3 years
* Passed Physical Activity Readiness Questionnaire + (PAR-Q+)
* Completed at an ACE baseline class
* Have access to a computer, laptop, iPad or Tablet with a video camera (with the Zoom app installed)
* Have access to an internet connection strong enough to support a live video broadcast

Exclusion Criteria:

* Active infections at the time of enrollment
* Enteral tube feeding/parenteral nutrition
* Mechanical or functional bowel obstruction due to any cause
* Cognitive impairment
* non-English speaking
* Neuromusculoskeletal issues that impede participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of Exercise Class Attendance (Cohort 1) | Beginning of exercise classes (week 1) until last day of exercise classes (week 8)
  Percentage of class attendance by all participants was assessed and deemed feasible if attendance was equal or above 70%.
Feasibility of Exercise Class Attendance (Cohort 2) | Beginning of exercise classes (week 1) until last day of exercise classes (week 12)
  Percentage of class attendance by all participants was assessed and deemed feasible if attendance was equal or above 70%.
Feasibility of Exercise Guidelines Adherence (Cohort 1) | Beginning of exercise classes (week 1) until last week of exercise classes (end of week 8)
  Percentage of participants meeting the exercise guidelines of 90 minutes of moderate to vigorous physical activity. 80% or higher adherence will be deemed feasible.
Feasibility of Exercise Guidelines Adherence (Cohort 2) | Beginning of exercise classes (week 1) until last week of exercise classes (end of week 12)
  Percentage of participants meeting the exercise guidelines of 90 minutes of moderate to vigorous physical activity. 80% or higher adherence will be deemed feasible.
Feasibility health coaching call completion (Cohort 1) | Beginning of exercise classes (week 1) until last week of exercise classes (week 8)
  Percentage of participants in the health coaching intervention completing all calls. 80% or higher completion will be deemed feasible.
Feasibility health coaching call completion (Cohort 2) | Beginning of exercise classes (week 1) until last week of exercise classes (week 12)
  Percentage of participants in the health coaching intervention completing all calls. 80% or higher completion will be deemed feasible.
Feasibility of Recruitment | Started about one month before study beginning and went until beginning of study (week 0)
  Percentage of participants signing up for the study over the eligible cancer survivors will be calculated. 50% or higher recruitment rate will be deemed feasible.
Fidelity of the health coaching intervention (Cohort 1) | Beginning of exercise classes (week 1) until last day of exercise classes (week 8)
  The fidelity of the health coaching intervention will be reported based on how close the intervention followed the protocol. Two sessions of each participant were randomly recorded (through envelope draw). After study completion a research assistant will analyze the recording with the health coaching protocol checklist. The research assistant will report percent agreement with the protocol (9 items for each health coaching session) and the time spent on each part of the health coaching call.
Fidelity of the health coaching intervention (Cohort 2) | Beginning of exercise classes (week 1) until last day of exercise classes (week 12)
  The fidelity of the health coaching intervention will be reported based on how close the intervention followed the protocol. Two sessions of each participant were randomly recorded (through envelope draw). After study completion a research assistant will analyze the recording with the health coaching protocol checklist. The research assistant will report percent agreement with the protocol (9 items for each health coaching session) and the time spent on each part of the health coaching call.
Fidelity of the exercise intervention (Cohort 1) | Beginning of exercise classes (week 1) until last day of exercise classes (week 8)
  The fidelity of the exercise intervention will be reported based on how close the intervention followed the protocol. The research coordinator joined each exercise class, reported on the class and compared the class structure to the exercise protocol checklist (4 items for each exercise class (including: Alterations to pre-class, warm-up, exercise circuits, cool-down, and post-class conversation)). Percent agreement between protocol and intervention across all classes will be reported. Additionally, the amount of times participants showed up late and the amount of times technical difficulties arose (including audio/video and log in complications) will be reported.
Fidelity of the exercise intervention (Cohort 2) | Beginning of exercise classes (week 1) until last day of exercise classes (week 12)
  The fidelity of the exercise intervention will be reported based on how close the intervention followed the protocol. The research coordinator joined each exercise class, reported on the class and compared the class structure to the exercise protocol checklist (4 items for each exercise class (including: Alterations to pre-class, warm-up, exercise circuits, cool-down, and post-class conversation)). Percent agreement between protocol and intervention across all classes will be reported. Additionally, the amount of times participants showed up late and the amount of times technical difficulties arose (including audio/video and log in complications) will be reported.
Feasibility of Study completion (Cohort 1) | Beginning of exercise classes (week 1) until last day of exercise classes (week 8)
  The attrition rate of the study was calculated as the percentage of dropouts out of all participants.
Feasibility of Study completion (Cohort 2) | Beginning of exercise classes (week 1) until last day of exercise classes (week 12)
  The attrition rate of the study was calculated as the percentage of dropouts out of all participants.
Feasibility of Assessment Completion (Questionnaire) (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Percentage of all assessments completed by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completion (Questionnaire) (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Percentage of all assessments completed by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completeness (Questionnaire) (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Percentage of all questions within the questionnaire answered by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completeness (Questionnaire) (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Percentage of all questions within the questionnaire answered by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completion (Physical functioning assessment) (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Percentage of all assessments completed by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completion (Physical functioning assessment) (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Percentage of all assessments completed by all participants was assessed and deemed feasible if completion was equal or above 70%.
Feasibility of Assessment Completion (Accelerometer) (Cohort 1) | Throughout the study from week 4 (due to COVID related delivery delays) until end of week 8
  Percentage of days accelerometer was worn as intended was assessed and deemed feasible if completed wear time days were equal or above 70% of overall study days. The accelerometer wearing time was calculated as following: a day was counted if the accelerometer was worn for more than 10 hours, the percentage of days worn over the overall days of the study was calculated.
Feasibility of Assessment Completion (Accelerometer) (Cohort 2) | Throughout the study from week 1 until end of week 12
  Percentage of days accelerometer was worn as intended was assessed and deemed feasible if completed wear time days were equal or above 70% of overall study days. The accelerometer wearing time was calculated as following: a day was counted if the accelerometer was worn for more than 10 hours, the percentage of days worn over the overall days of the study was calculated.
Semi-Structured Interview (Feasibility) | Post-intervention (week 9 (first wave) or week 13 (second wave))
  Include participant satisfaction, barrier management, pros/cons to the home-setting, value of the health coaching support, and facilitators to maintaining PA levels.

SECONDARY OUTCOMES:
Physical Activity Minutes Per Week (objective) (Cohort 1) | Throughout the study from week 4 (due to COVID related delivery delays) until end of week 8
  Change in activity levels from pre to post; Number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate to vigorous intensity exercise, based on accelerometer data from commercially-available activity tracker.
  For the activity tracker each minute in the 55-70% age predicted HRmax will be evaluated as moderate intensity and above 70% of HRmax will be evaluated as vigorous intensity.
  Vigorous intensity minutes of physical activity will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes.
Physical Activity Minutes Per Week (objective) (Cohort 2) | Throughout the study from week 1 until end of week 12
  Change in activity levels from pre to post; Number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate to vigorous intensity exercise, based on accelerometer data from commercially-available activity tracker.
  For the activity tracker each minute in the 55-70% age predicted HRmax will be evaluated as moderate intensity and above 70% of HRmax will be evaluated as vigorous intensity.
  Vigorous intensity minutes of physical activity will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes.
Physical Activity Minutes Per Week (subjective) (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in activity levels from pre to post; Number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate to vigorous intensity exercise, based on the modified Godin Leisure Time Exercise Questionnaire (mGLTEQ).
  In the mGLTEQ all dimensions (strenuous exercise, moderate exercise, mild exercise, resistance training, and flexibility) will be looked at separately and weekly minutes will be calculated by multiplying duration times frequency of sessions.
  Vigorous intensity minutes of physical activity will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes.
Physical Activity Minutes Per Week (subjective) (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in activity levels from pre to post; Number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate to vigorous intensity exercise, based on the modified Godin Leisure Time Exercise Questionnaire (mGLTEQ).
  In the mGLTEQ all dimensions (strenuous exercise, moderate exercise, mild exercise, resistance training, and flexibility) will be looked at separately and weekly minutes will be calculated by multiplying duration times frequency of sessions.
  Vigorous intensity minutes of physical activity will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes.
Body Composition (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in body mass index (BMI)
Body Composition (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in body mass index (BMI)
Aerobic Endurance (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in 2 minute step test (steps) results
Aerobic Endurance (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in 2 minute step test (steps) results
Strength Endurance (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in sit-to-stand (number of repetitions in 30 seconds)
Strength Endurance (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in sit-to-stand (number of repetitions in 30 seconds)
Upper extremity flexibility (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in active shoulder flexion range of motion (degrees)
Upper extremity flexibility (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in active shoulder flexion range of motion (degrees)
Lower extremity flexibility (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in sit-and-reach test (cm)
Lower extremity flexibility (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in sit-and-reach test (cm)
Balance (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in one legged stance test (seconds)
Balance (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in one legged stance test (seconds)
Barrier Self-Efficacy (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in barrier self-efficacy measured by Rogers et al 9 item scale (0-100).
Barrier Self-Efficacy (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in barrier self-efficacy measured by Rogers et al 9 item scale (0-100).
General Wellbeing (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in overall Functional Assessment of Cancer Therapy - General subscale (FACT-G) score as well as the single domains (Physical Well-being, Social/Family Well-being, Emotional Well-being, Functional Well-being)
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much"
General Wellbeing (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in overall Functional Assessment of Cancer Therapy - General subscale (FACT-G) score as well as the single domains (Physical Well-being, Social/Family Well-being, Emotional Well-being, Functional Well-being)
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much"
Fatigue (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in the overall Functional Assessment of Chronic Illness Therapy - Fatigue subscale (FACIT-F) score
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
Fatigue (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in the overall Functional Assessment of Chronic Illness Therapy - Fatigue subscale (FACIT-F) score
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
Social Support (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in the Oslo Social Support Scale (OSSS-3) score
Social Support (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in the Oslo Social Support Scale (OSSS-3) score
Loneliness (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in the UCLA Loneliness Scale Short Version (ULS-6) score
Loneliness (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in the UCLA Loneliness Scale Short Version (ULS-6) score
Stress (Cohort 1) | Before study (week 0) and after study completion (Week 9)
  Change in the Perceived Stress Scale (PSS) score
Stress (Cohort 2) | Before study (week 0) and after study completion (Week 13)
  Change in the Perceived Stress Scale (PSS) score
Garmin Activity Tracker Usage (Cohort 2) | Post-intervention (week 13)
  Participants were asked how frequently they used the following features on the Garmin Vivosmart4: Steps, Floors climbed, Activity Tracking, Intensity minutes tracking, Heart Rate tracking, Sleep monitoring, Stress monitoring, Body battery, and Calories burned. The answer options for the use of each Garmin function were: Never, Once, Twice, Once every two weeks, Once a week, twice a week, almost every day, every day, or multiple times a day.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Faculty of Kinesiology University of Calgary, Calgary, Alberta
  - Health and Wellness Lab, University of Calgary, Calgary, Alberta

REFERENCES:
- [Derived] Eisele M, Pohl AJ, McDonough MH, McNeely ML, Ester M, Daun JT, Twomey R, Culos-Reed SN. The online delivery of exercise oncology classes supported with health coaching: a parallel pilot randomized controlled trial. Pilot Feasibility Stud. 2023 May 12;9(1):82. doi: 10.1186/s40814-023-01316-z. PMID 37173764